CLINICAL TRIAL: NCT00883987
Title: A Pilot Project to Study the Effect of Four Osteopathic Treatments on Trunk Muscle Firing Patterns and Temporospatial Parameters of Gait in Persons With Chronic Low Back Pain
Brief Title: Osteopathic Treatment of Low Back Pain
Status: Completed | Type: Observational
Sponsor: Mary Lynch (Other)
Responsible Party: Sponsor-Investigator, Mary Lynch, MD FRCPC, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Other Study IDs: CDHA-RS/2009-366
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Back Pain: Patients with chronic mechanical low back pain (Chronic low back pain is defined as having "pain between the lower ribs and gluteal folds, with minimal radiation to the thigh and never below the knee, present for a minimum of seven weeks")

SUMMARY:
Eighty percent of Canadians experience low back pain (LBP) at some point in their life (Waddell, 1987), with a point prevalence of up to 30 percent (O'Sullivan, 2005; Waddell, 1987). Low back pain has severe economic ramifications. Most incidents of low back pain occur during the prime working years of life, with an estimated cost to the economy at $14,744 Canadian dollars per person per year (Health Canada, 1998). Indirect costs in the form of long-term disability were highest for disorders of arthritis and chronic back pain (Health Canada, 1998). It has been estimated that 12 percent of patients will experience disability within one year after their first episode of low back pain (Banner, 2006). Evidence based diagnosis and treatment is important for desirable outcomes.

The investigators predict that there will be changes in A) trunk muscle electromyographic patterns and in temporo-spatial gait patterns following osteopathic treatment.

DETAILED DESCRIPTION:
Research has outlined trunk muscle activation patterns in patients with LBP are different from those who do not suffer from low back pain (Clarke-Davidson and Hubley-Kozey, 2005; Hodges, 1996 and 1997; McGill, 2001 and 2002). Osteopathic research has documented the effects of osteopathic manipulative therapy (OMT) on EMG activity in patients with low back pain (Beckman, Harrington, Dostert, et al., 1991; Ellestad, Nagle, Boesler, et al.,1988; Krpan, Harrington, Beckman, 1992; Steiner, Park, Guzels, 1991) however these studies were limited in design and methodology.

In a controlled trial which measured levels of cellular enzymes to monitor tissue damage during OMT, blood serum enzyme levels did not change as a result of manipulation. More important, EMG levels decreased. OMT did not damage tissue but changed motor neuron activity (Rowane, Horner, Warner, et al., 1989). Beckman, et al., (1991) observed a reduction in EMG activity following OMT in patients with low back pain and found increased skin blood flow as measured by laser doppler flow meter. Steiner et al. (1991), reveal reduction to muscle spasm as measured by EMG in patients with low back pain following OMT. A further study (Ellestad, et al., 1988) noted decreased EMG activity during motion in patients with chronic low back pain. Thus there is preliminary work providing support for reduced EMG activity following OMT within low back pain treatment groups. However there is a need for further research in this area.

We also want to determine the role of manual therapy (osteopathy) in the management of gait dysfunction in this patient population. Patients with LBP present with reduced gait speed, poor thoraco-pelvic coordination and increased erector spinae activity (Lamoth et al. 2002 and 2006), altered weight bearing (Ellen Lee et al., 2007) and reduced single leg stance balance in static conditions (Louto et al., 1998).

Reduced thoraco-pelvic coordination leads to muscular stabilizing effects, altered kinematics, trunk rigidity, and reduced walking velocity (Lamoth et al., 2002). Specific impairments of body structure and function can reduce gait speed in older adults (Kerrigan, Todd, Della Cruce, 1998). Osteopathic intervention targets movement impairments of body structure and should change gait speed in patients with chronic LBP. Mal-alignment contributes to pathology in the pelvis and lumbar spine which can lead to degenerative changes, instability and pain (Aebi, 2005; Gurney, 2002; Steinburg, Luger, Arbel, et al., 2003). The focus of osteopathy is to restore mobility and alignment throughout the whole kinetic chain (Kutchera and Kutchera, 1991; Seffinger, 2007).

Improvement in gait speed and joint motion is shown after mobilization exercises to the ankle and hip in the elderly (Christiansen, 2003). A kinetic relationship links the ankle and pelvis (Gurney, 2002; Khamis & Yizhar, 2007; Pinto, Souza, Tede, et al., 2008). Cephalo-caudal (pelvis affects ankle), caudal-cephalo (ankle affects pelvis) and ipsilateral-contralateral (one leg affects the other via the pelvis) alignment and kinematic relationships occur when lower extremity joints are maintained in altered positions (Pinto, et al., 2008). Can movement dysfunction secondary to impaired mobility and mal-alignment contribute to pain and antalgic gait?

ELIGIBILITY:
Inclusion Criteria:

* between the age of 19 and 55 years old,
* able to walk without assistance and /or assistive devices at least 4.7 meters.
* have adequate hearing acuity to detect verbal instructions.
* have adequate visual acuity to walk safely in usual ambient lighting without holding onto objects.
* be able to speak and comprehend English,
* have sufficient cognitive ability to follow instructions, and to provide informed consent, as defined by a Mini Mental Status Examination score of greater than 23 out of 30, performed by the research coordinator.

Exclusion Criteria:

* have had neurological signs and symptoms, or complications such as tumor or infection.
* are active in a claim pertaining to a motor vehicle accident or work injury or under any litigation for their pain.
* have had previous osteopathic treatment in the last year.
* had more than one abdominal surgery, or spinal fracture, or structural deformity such as scoliosis or spondylolithesis (Hubley-Kozey, 2002)
* have severe cardiopulmonary disease as determined by a health questionnaire with symptoms such as shortness of breath or chest pain on mild exertion or at rest,
* history of severe neurological disorder that impairs balance and mobility eg stroke, Parkinson's disease, peripheral neuropathy
* have pain that leads to severe discomfort with minimal movement,
* have significant musculoskeletal impairment e.g. arthritis that leads to severe discomfort with walking that could lead to an abnormal gait,
* have cognitive compromise impairing ability to care for oneself, and ability to provide informed consent,
* have dizziness while standing,
* have a history of falls in previous month that might make it unsafe to participate in a gait study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with chronic mechanical low back pain (Chronic low back pain is defined as having "pain between the lower ribs and gluteal folds, with minimal radiation to the thigh and never below the knee, present for a minimum of seven weeks"
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Two primary outcome measures will be used for this study. The GAITRite gait analysis system and surface electromyography (EMG) respectively. | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lynch, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- CDHA Pain Management Unit, Halifax, Nova Scotia, Canada